CLINICAL TRIAL: NCT03586297
Title: Gut and Intratumoral Microbiome Effect on the Neoadjuvant Chemotherapy-induced Immunosurveillance in Triple Negative Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: BCRF 2017; PRO2017-0331 (Other: HackensackUMC)
Record Dates: First submitted 2018-06-11; First posted 2018-07-13 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Triple Negative Breast Cancer
Keywords: BCRF; Microbiome; Intratumoal microbiota
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and Blood Specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The probability of pCR in TNBC patients receiving standard of care neoadjuvant chemotherapy treatment is associated with the dominance of specific intestinal and intratumoral microbiota that promote anti-tumor immunosurveillance.

DETAILED DESCRIPTION:
This is a prospective study of newly diagnosed triple negative breast cancer (TNBC) patients undergoing standard of care neoadjuvant chemotherapy and correlate gut and intratumoral microbiome composition and anti-tumor immune responses with pCR.

The biopsy at diagnosis will be used as a pretreatment control for the assessment of TILs, PD-L1 expression, immune signature profiles. Both tumor and "normal" adjacent non-tumor tissue will be evaluated. Stool and peripheral blood (PB) samples will be collected at time of consent for therapy. TNBC patients will be treated with the standard of care neoadjuvant chemotherapy. At mid-treatment (MT), an elective tumor biopsy will be performed and stool and PB samples will be collected. At time of surgery, after the completion of neoadjuvant chemotherapy (at the discretion of the medical oncologist), resected tumor and "normal" adjacent non-tumor tissue, stool and PB samples will be collected.

Pre- , mid- and post-therapy immune phenotyping/profiling will be determined in PB samples and patient biopsies. The overall composition of the gut microbiome will also be determined in patient stool samples.

The overview of the study is presented below:

1. Regimen and duration of neoadjuvant chemotherapy is at the discretion of the medical oncologist.
2. Cycle 1 refers to first dose of each treatment.
3. Tumor morphology, IHC and FISH will be performed at diagnosis of TNBC. Criteria for newly diagnosed TNBC: <1% of ER and PR immunoreactivity and HER2- by FISH or IHC staining 0 or 1+ and T1 (T1: <1.5 cm) mass lesion or greater.
4. For correlative studies, collection of PB will be at day 1 of cycle 1, day 1 of cycle 1 of T and end of treatment, prior to surgery. Eight 8x tubes, seven (7) yellow top tubes (BD Vacutainer ACD Solution A Blood Collection tubes - 8.5ml) and one (1) Streck tube . Immunophenotying, gene expression profiling and assessment of cytokine/chemokine and other mediators production will be performed.
5. For correlative studies, Stool collection will be collected up to 48 hours prior to drug administration on day 1 of cycle 1 and day of surgery. Sequencing of the gut and intratumoral microbiome and gene-associated pathways will be performed by 16S rRNA and shotgun metagenomics sequencing.
6. For correlative studies, immunostaining of fixed tissue for PD-L1 or other immune marker expression on tumor cells and for the in situ presence of various T cell subset markers with PD1 expression will be performed. Isolation of DNA and RNA will be performed from formalin-fixed tissues.
7. Tumor biopsy for mid-treatment (MT). This biopsy will be offered and performed upon consent of patient.
8. This tissue will be provided by Pathology Department upon processing of surgical specimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed new diagnosis of TNBC (<5% of ER and PR immunoreactivity and HER2- by FISH or IHC staining 0 or 1+)
* >18 years
* 1.5 cm mass lesion or greater
* Tumor amenable to percutaneous core biopsy

Exclusion Criteria:

* chronic anticoagulation therapy
* prior ipsilateral breast surgery, ipsilateral radiotherapy, hormonal therapy or systemic chemotherapy
* Prolonged antibiotic treatment > 10 days within 1 month of neoadjuvant chemotherapy as prevention or suppression of an ongoing infection
* lactating
* pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be Female
Study Population: Newly Diagnosed Triple Negative Breast Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-08-27 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response | completion of chemotherapy, approximately 18 weeks.
  The primary objective of this study is to determine if the probability of pCR (pathologic complete response) in TNBC (triple negative breast cancer) patients treated with standard of care neoadjuvant chemotherapy is correlated with variability in the composition of intestinal and intratumoral microbiota and subsequent short-term alterations in that composition.

SECONDARY OUTCOMES:
Other Correlations between Pathologic complete Response | completion of chemotherapy, approximately 18 weeks.
  Determine whether the correlation between specific microbiota and the probability of pCR is predictive for the resolution of T cell exhaustion.
Other Correlations between Pathologic complete Response | completion of chemotherapy, approximately 18 weeks.
  Determine if specific microbiota correlated with the probability of pCR are associated with the anti-tumor innate and adaptive immune responses in the tumor site and peripheral blood.
Other Correlations between Pathologic complete Response | completion of chemotherapy, approximately 18 weeks.
  Determine the predictive values of baseline tumor PD-L1 (Programmed death-ligand 1) expression and PD-1 and other immune checkpoint inhibitory markers in TILs (tumor infiltrating lymphocytes) with pCR.

CONTACTS AND LOCATIONS:
Overall Officials: Marson Davidson, MD, Principal Investigator — Hackensack Meridian Health
Locations (3):
- United States (3):
  - Yale University - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Hackensack Meridian Health, Hackensack, New Jersey